CLINICAL TRIAL: NCT03292874
Title: Evaluation of a Novel High-Resolution Diffusion-Weighted MRI Sequence
Brief Title: High Resolution MRI Study for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Hyung L. Kim, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00049177
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, paired imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Paired imaging (Other): Single arm, paired imaging of high resolution MRI (hrMRI) and stand MRI (sMRI)
  Interventions: Diagnostic Test: high resolution MRI (hrMRI)

INTERVENTIONS:
Diagnostic Test: high resolution MRI (hrMRI) — high resolution MRI (hrMRI) and standard MRI (sMRI) will be obtained at baseline and again in approximately 1 year in patients on prostate cancer active surveillance.

SUMMARY:
This high resolution MRI (hrMRI), along with stand MRI (sMRI) will be obtained at baseline and again in approximately 1 year in patients on prostate cancer active surveillance. Changes in lesion size and ADC values will be assessed on the serial studies. This study evaluates the hypothesis that hrMRI will detect changes that sMRI cannot detect and that these changes will correlate with prostate cancer progression as determined on prostate biopsy.

DETAILED DESCRIPTION:
2.0 BACKGROUND AND RATIONALE

Multiparametric MRI Multiparametric MRI combining T2-weighted, diffusion-weighted, and dynamic contrast enhanced (DCE) images is commonly employed for detection and localization of prostate lesions. Diffusion-weighted imaging (DWI) is sensitive to the diffusion of water molecules interacting with surrounding macromolecules. DWI, which provides a quantitative biological parameter called apparent diffusion coefficient (ADC) value, is a robust MRI parameter for differentiating benign and malignant prostate tissue. In fact, the latest version of the Prostate Imaging-Reporting and Data System (PI-RADS) scoring system relies almost exclusively on DWI to identify tumors in the peripheral zone, which is where the vast majority of prostate cancers form. Findings on T2 images are not used to identify cancer, and DCE images are only used to differentiate between some PI-RADS 3 and 4 lesions. In a pilot study of prostate cancer AS, DW-MRI was useful for detecting progression of Gleason score based on changes in ADC value. Tumor size is another important clinical criterion for defining low risk prostate cancer, and tumor size based on DWI has been shown to crudely predict low risk prostate cancer. However, conventional DWI using single-shot echo-planar imaging is unable to detect small tumors, low grade tumors, or small changes in tumor size on serial imaging. Approximately 20% of small, low grade tumors found in men on AS are detected on modern prostate MRI.

High Resolution MRI Investigators introduce a new three-dimensional (3D) high-resolution diffusion-weighted imaging sequence (HR-DWI), which improves image quality while conferring at least a 5-fold improvement in resolution when compared to standard two-dimensional (2D) DWI (S-DWI). This novel 3D DWI technique has been developed by our team and can be applied on existing 1.5T or 3T MRI systems. S-DWI suffers from two important limitations. a) It uses single-shot echo-planar imaging (EPI) for data acquisition, which produces magnetic susceptibility induced streaking artifacts and geometric distortions so that round objects may appear oval. b) The relatively low signal-to-noise ratio and 2D image acquisition with S-DWI limit spatial resolution, which is defined by the minimum distance between two objects required to resolve them uniquely. Our HR-DWI overcomes these limitations by using magnetization prepared, multi-shot, turbo-spin-echo acquisition, which improves signal-to-noise ratio (SNR), spatial resolution, and image quality, and eliminates geometric distortions and streaking artifacts associated with EPI.

Preliminary studies

In preliminary studies assessing the performance of our HR-DWI in a prospective pilot trial of prostate cancer AS patients, the technique could detect tumors not seen on S-DWI and measure ADC, which correlates with grade. This is important because the long-term natural history of small prostate cancers invisible to S-DWI has never been prospectively defined, in part due to lack of adequate imaging technology. In the era of molecular diagnostics and next-generation sequencing, an important step in understanding the biology of these lesions is to develop technologies to image and characterize these lesions. Importance of HR-DWI includes:

* Better imaging will allow these lesions to be monitored serially and targeted for biopsy, providing tissue for both histologic and molecular characterization.
* Higher resolution imaging will better delineate tumor boundaries, which can improve tumor staging and identify margins during partial-gland ablation by cryotherapy or high intensity focused ultrasound (HIFU), which was approved in 2015 by the U.S. FDA.
* Improved imaging resolution will allow for more accurate measurement of tumor size and ADC, and detection of small changes in size or grade over time. Standard prostate DWI has poor resolution; therefore, tumor growth kinetics have never been accepted as clinical criteria for cancer progression while on AS. If tumor growth kinetics or changes in grade determined by ADC prove prognostic, AS can rely less on serial transrectal biopsies, which can lead to serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients diagnosed with clinically localized prostate cancer
* Low or Low-intermediate Risk Prostate cancer1 defined as:
* Pre-operative prostate specific antigen (PSA) ≤ 20.0 ng/ml
* Clinical stage cT1 or cT2
* Gleason score 3+3 or 3+4
* Patients choosing AS or already on AS as primary management strategy
* No previous treatment for prostate cancer with radiotherapy, chemotherapy, or hormonal therapy
* No contraindications for gadolinium enhanced MRI

Exclusion Criteria:

* No exclusion criteria

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyung L Kim, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paired Imaging: Single arm, paired imaging of high resolution MRI (hrMRI) and standard MRI (sMRI)
  high resolution MRI (hrMRI): high resolution MRI (hrMRI) and standard MRI (sMRI) will be obtained at baseline and again in approximately 1 year in patients on prostate cancer active surveillance.
Period: Overall Study
Arm/Group | Paired Imaging
Started | 64
Completed | 59
Not Completed | 5
Not completed — Due to pandemic | 5

BASELINE CHARACTERISTICS:
Arm/Group | Paired Imaging
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
PSA [Mean (Standard Deviation); unit: nanograms per milliliter] | 6.0 (2.8)
Histologic Grade [Count of Participants; unit: Participants] — Histologic grade from prostate biopsy
  Participants
    Low grade (Gleason 3+3) | 45
    Intermediate grade (Gleason 3+4) | 14
No. positive cores on prostate biopsy [Mean (Standard Deviation); unit: Number of positive cores] — Number of positive cores per patient on a standard prostate biopsy involving systematic sampling of the prostate.
  Number of positive cores | 2.9 (2.4)
No. prior biopsies [Count of Participants; unit: Participants]
  0 | 41
  1 | 8
  >1 | 10
Stage [Count of Participants; unit: Participants] — Determined from digital rectal exam of the prostate
  Participants
    T1c (non-palpable tumor) | 58
    T2a (palpable tumor) | 1

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of High Resolution Versus Standard MRI in Identifying Adverse Histology
Description: The primary endpoint of the clinical trial was the presence of adverse histology (AH) on prostate biopsy. We defined adverse histology (AH) as either overall Gleason score of 7 or more on any biopsy, or an increase of 3 or more positive cores on serial systematic biopsies. The primary hypothesis was that change in tumor size or apparent diffusion coefficient (ADC) as detected by high resolution MRI (hrMRI) would better predict AH than standard MRI (sMRI). AH histology was a measure intended to capture patients with high Gleason grade component (i.e. Gleason Grade 4 or 5) and patients progressing (e.g. from Gleason Group 1 to Gleason Group 2 or from Gleason Group 2 to Gleason Group 3). The sample size was too small and the followup duration of approximately 12 months was too short to assess only true cancer progression as the endpoint. The presence of AH alone is clinically important since these patients may need close followup and may consider definitive local therapy.
Time Frame: 6-12 months after enrollment
Population: Each participant underwent both sMRI and hrMRI.
Measure: Number; unit: percent
Groups:
- High Resolution MRI (hrMRI); Standard MRI (sMRI): All patients underwent hrMRI and sMRI.
Arm/Group | High Resolution MRI (hrMRI) | Standard MRI (sMRI)
Number analyzed (Participants) | 59 | 59
percent
  sensitivity | 75 | 71
  specificity | 84 | 54.8

2. Primary Outcome: Area Under the Receiver Operator Curve of High Resolution Versus Standard MRI in Identifying Adverse Histology
Description: as for outcome 1
Time Frame: 6-12 months after enrollment
Population: Each participant underwent both sMRI and hrMRI. Each was assess for predicting AH.
Measure: Number; unit: probability
Arm/Group | High Resolution MRI (hrMRI) | Standard MRI (sMRI)
Number analyzed (Participants) | 59 | 59
probability | 0.794 | 0.631
Statistical Analysis 1: Comparison: High Resolution MRI (hrMRI) vs Standard MRI (sMRI); Test type: Superiority; p = 0.014, nonparametric method — Areas under the receiver operating characteristics curve (AUC) were compared between models with standard and high-resolution MRI variables using the nonparametric method described by DeLong. DeLong. Biometrics 1988;44(3):837-45

ADVERSE EVENTS:
Time Frame: 12 months
Description: This is an imaging study of a novel MRI.
Groups:
- hrMRI: high resolution MRI
- sMRI: standard MRI
Arm/Group | hrMRI | sMRI
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

LIMITATIONS AND CAVEATS:
The number of patients in our study was relatively small. The reference standard was prostate biopsies, which is subject to sampling error. However, this was necessary when investigating a low-risk, small-volume cancer that is managed nonoperatively. Our study was performed at a single center and the imaging protocol was developed by our team.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03292874/Prot_SAP_000.pdf